CLINICAL TRIAL: NCT04062253
Title: Addressing the Cascade of Care in Vulnerable Populations With Poor Access to Healthcare in Madrid
Acronym: (UMC)
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Principal Investigator, Pablo Ryan, Principal Investigator, Hospital Universitario Infanta Leonor
Other Study IDs: 19/05
Record Dates: First submitted 2019-05-10; First posted 2019-08-20 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: HCV Infection; HIV Infections; Drug Use; HBV (Hepatitis B Virus); Viral Hepatitis
Keywords: HIV; HCV; PWID (Persons who inject drugs); Screening; Diagnosis; Linkage to care; Treatment
MeSH Terms: conditions — Hepatitis C; HIV Infections; Hepatitis B; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCV or HIV negative: Individuals who test negative for HCV or HIV are given information regarding ways of transmission.
  Interventions: Diagnostic Test: HCV rapid test
- HCV and HIV positive: Individuals with a positive test for HCV o HIV are offered delivery or accompaniment to specialist health care.
  Interventions: Diagnostic Test: HCV rapid test

INTERVENTIONS:
Diagnostic Test: HCV rapid test — Individuals who test positive for either HIV or HCV are offered PCR (polymerase chain reaction) testing with the xpert technology. Patients with a confirmed active infection are offered delivery and are taken into hospital.
  Other Names: HIV rapid test; Xpert HCV viral load; Xpert HIV viral load; Linkage to care

SUMMARY:
Data on the prevalence of hepatitis C virus (HCV) for other vulnerable groups in Madrid, such as homeless persons and migrants, are scarce, and it is now necessary to implement intervention and elimination plans.

Vulnerable groups have poor access to healthcare and are therefore not systematically screened for HCV. On the occasions they are shown to be positive, subsequent follow-up in the health system and the possibility of cure are poor.

The use of a mobile unit to approach vulnerable populations is essential for better characterization of risk behaviors and of the magnitude of HCV. The integration of healthcare personnel in mobile units enables counseling on prevention and intervention when needed.

Primary objective Evaluate the impact of the HCV care cascade on vulnerable populations who gather at hot spots in Madrid (shantytowns, homeless shelters and places were street prostitution is practiced) by means of a multilevel outreach project.

SURVEILLANCE:

Active screening for HCV among vulnerable individuals in populations with a high prevalence of HCV will be carried out in hot spots in Madrid, namely, Cañada Real shanty town, mobile harm reduction units, institutions providing social assistance, public areas, homeless shelters and places where street prostitution is practiced. An agreement with the Madrid Council (MCC) is under way to provide social centers for HCV screening.

A mobile unit will approach the hot spots following a predefined schedule. The mobile unit consists of a van adapted for the project and a car. HCV screening of vulnerable individuals will be performed by a nurse and an educator hired specifically for that purpose.

Active HCV screening and prevention in vulnerable individuals should be a priority and a responsibility shared by both the MCC and the SERMAS (Servicio Madridleño de Salud). The investigators plan to establish an agreement with public health authorities to give continuity to this project and to carry out proactive HCV screening through integration with various centers and networks dependent on the MCC and SERMAS.

The project will establish the foundations of integrated cooperation between an HCV clinic in a hospital setting and harm reduction units and other resources and networks dependent on the institutions mentioned above. As has been observed with other interventions, the functional objective of this project is to provide continuity of care from the institutions.

Study Duration (in months) 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Vulnerable populations who include one or more of the following:

  * Persons who inject drugs,
  * Homeless,
  * Migrants
  * Sex workers

Exclusion Criteria:

* Not signing inform consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons who inject drugs (PWID), homeless people, migrants and sex workers are vulnerable populations that have a high prevalence of active hepatitis C virus (HCV) infection. According to local data, the prevalence of HCV in drug users ranges from 20% to 60%, depending on whether they inject drugs or not. Data on the HCV prevalence for the other vulnerable groups (homeless, migrants…) in Madrid is scarce and necessary to implement intervention and elimination plans.
Sampling Method: Non-Probability Sample
Enrollment: 2001 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who have a positive RNA HCV test | 1 year
  Percentage of those participants screened for HCV, Who hace a positive RNA HCV test using a Genexpret test onsite.
Percentage of Participants Who have a positive HIV rapid test | 1 year
  Percentage of those participants screened for HIV, Who hace a positive test

SECONDARY OUTCOMES:
Percentage of Participants Who have an active HCV infection and start HCV therapy. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Unidad Movil de Cribado, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Itineraries and schedules of the project. — http://unidadmovil.es